CLINICAL TRIAL: NCT00759772
Title: The Role of PTH in Low Bone Mass in Anorexia Nervosa
Brief Title: The Role of Parathyroid Hormone (PTH) in Low Bone Mass in Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Pouneh K. Fazeli, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 829
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Anorexia Nervosa; Osteoporosis
Keywords: Anorexia Nervosa; Disordered Eating; Osteoporosis; Parathyroid Hormone; Bone
MeSH Terms: conditions — Anorexia Nervosa; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Active Comparator)
  Interventions: Drug: Teriparatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — sc daily for 6 months
  Arms: Placebo
Drug: Teriparatide — 20 mcg sc daily for 6 months
  Arms: Teriparatide

SUMMARY:
Decreased bone strength is a common and serious medical problem present in many women with anorexia nervosa, or disordered eating. Women with decreased bone strength are more likely to suffer broken bones than women with normal bone strength.

We are investigating whether a hormone that is naturally produced by the human body -- parathyroid hormone (PTH) -- can help strengthen the bones of women with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia Nervosa affects 0.5-1% of college-age women in the US and is associated with a number of significant medical conditions including bone loss. A majority of women with anorexia nervosa have bone loss and 50% have bone mineral density measurements greater than 2 standard deviations below normative means. Bone loss in anorexia nervosa is characterized by a decrease in bone formation, therefore therapy with an anabolic agent may be an effective treatment approach. In a randomized, single-blinded, placebo-controlled trial, we will study the effects of parathyroid hormone on low bone mass in anorexia nervosa, specifically looking at the effects of parathyroid hormone on bone mineral density (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa
* Women, age 30-70 years
* Osteoporosis or history of clinical fractures (spine, wrist, hip or ribs)

Exclusion Criteria:

* Diseases known to affect bone metabolism
* Hyperparathyroidism
* Medications known to affect bone metabolism in last 12 weeks (or bisphosphonate use in last 1 year)
* Pregnant and/or breastfeeding
* Diabetes mellitus
* History of malignancy involving or affecting the bone, any active malignancy, and/or radiation therapy to the bone
* Fractures of a bone other than a finger or toe in last 1 year

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pouneh K Fazeli, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Teriparatide: Teriparatide 20 mcg sc daily for 6 months
- Placebo: Placebo: Placebo 20 mcg sc daily for 6 months
Period: Overall Study
Arm/Group | Teriparatide | Placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.6) | 47.1 (7.6) | 47.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lumbar Spine Bone Mineral Density
Description: Percent increase or decrease in lumbar spine bone mineral density between baseline and 6 months (treatment period)
Time Frame: Baseline and 6 months
Population: All participants were included in analysis (intention to treat).
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 12 | 11
percentage of change | 5.6 (1.3) | 0.2 (0.7)
Statistical Analysis 1: Comparison: Teriparatide vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — Calculated p-value

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were monitored/assessed without regard to the specific Adverse Event Term. Adverse event descriptions are listed in the table.
Arm/Group | Teriparatide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/11
Other Adverse Events (participants affected / at risk) | 12/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide (N=12) | Placebo (N=11)
Hospitalization or exacerbation (Psychiatric disorders) | 2 | 3 — Subjects hospitalized (or had worsening of) anorexia nervosa-related complications (all were considered unrelated to study drug)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide (N=12) | Placebo (N=12)
Lightheadedness (Nervous system disorders) | 4 | 6
Muscle pain/spasm (Musculoskeletal and connective tissue disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 1 | 3
Headache (Nervous system disorders) | 6 | 5
Injection site ecchymoses, bruising, erythema (Skin and subcutaneous tissue disorders) | 8 | 9
Elevated serum calcium (Endocrine disorders) | 3 | 0
Elevated 24hr urine calcium (Endocrine disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No